CLINICAL TRIAL: NCT03730155
Title: Compassion Cultivation Training (CCT): A Preventive Intervention for Caregivers of People Who Suffer From a Mental Illness
Brief Title: Compassion Cultivation Training (CCT): An Intervention for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Compassion2018
Record Dates: First submitted 2018-10-24; First posted 2018-11-05 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2018-10

CONDITIONS: Psychological Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCT intervention (Experimental): CCT intervention. 8 weeks with 2 hours session every week. Homework approx. 25 min. of meditation daily.
  Interventions: Other: CCT intervention.
- Control waitlist (No Intervention): No treatment given. Participants only answer questionnaire packages.

INTERVENTIONS:
Other: CCT intervention. — 8-week course with 2 hours sessions weekly. Participants should meditate 25 min. pr. day during the 8 weeks.
  Arms: CCT intervention

SUMMARY:
This study will begin a novel line of research on CCT in Denmark as a preventive intervention for caregivers of people suffering from a mental illness. The primary aim of the study is to investigate the effectiveness of a Compassion Cultivation Training (CCT) course on psychological distress of informal caregivers.

DETAILED DESCRIPTION:
Hypothesis 1: It is hypothesized that caregivers in CCT will reduce psychological distress, relative to control participants, as measured by the Depression Anxiety Stress Scale (DASS) at baseline (T0), post intervention (T1), 3-month (T2) and 6-month (T3).

Hypothesis 2: It is hypothesized that caregivers in CCT, relative to control participants, will increase compassion for self and others, show greater acceptance of difficult emotions and decrease emotion suppression as measured by Self-Compassion Scale Short Form (SCS-12), Multidimensional Compassion Scale (MCS), Perceived Stress Scale, (PSS), The Emotion Regulation Questionnaire (ERQ)), The Five Facet Mindfulness Questionnaire (FFMQ-15), Brief Resilience Scale (BRS) and WHO-5 measured at T0, T1, T2, and T3.

Hypothesis of Mechanisms: Improvements on these skills will mediate the effects of treatment and outcome. Specifically: a) increase in compassion for self and others (SCS-12 and MCS) will mediate the effects of emotion regulation skills (i.e. greater acceptance of difficult emotions and therefore less suppression of difficult emotions) and b) increase in emotion regulation skills (ERQ) (i.e. greater acceptance of difficult emotions and therefore less suppression of difficult emotions) will mediate the effects of psychological distress (DASS) in informal caregivers.

Methods Research design The effect of CCT will be evaluated in a parallel randomised controlled trial including 77 participants in the intervention group and 77 in a wait-list group.

Participants will be recruited through primary care physicians. The Danish Center for Mindfulness, Aarhus University has a good history of recruiting participants for their trials, due to well established relationships primary care physicians. Recruitment will also be carried out in collaboration with the national association for caregivers; Bedre Psykiatri, Landsforeningen for pårørende (Better Psychiatry, national association for caregivers), through Psykiatrifonden (The Danish Mental Health Fund), who acknowledge and support this research as they are keenly aware of the great need for interventions for informal caregivers. Lastly, we will recruit through social media such as Facebook, Twitter, and the Danish Center for Mindfulness website. Randomization After informed consent and T (0) measures, participants will be randomized to either CCT (N=77) or waitlist control group (N=77) using a computer algorithm with predefined, concealed random numbers. An independent statistician will manage the randomization by giving all registered participants either a number of "1" or "2" in sequence. The participants with "1" will be assigned to the immediate intervention group and those with "2" to a waitlist control group. We will not use "treatment" or "control" group to mention the allocation. All subjects will be told that they will be arranged into two groups to attend the CCT session separately due to resource limitations. The independent clinical assistant will call participants to let them know the group they belong to, either the immediate group or the waitlist group.

Procedure Eligible participants, meeting all study criteria, are asked to participate in the Randomized Controlled Trail (RCT). All participants will be given psychological, and demographic measurements at baseline (T0), and psychological measures at post intervention (T1), 3-month follow-up (T2) and 6-month follow-up (T3), The study will be registered in ClinicalTrails.gov before commencement. The investigators will specifically ask that the participants in the waitlist control group do not start any other intervention during the study period.

Data Collection Eligible participants will receive an email with a link to the measurements that must be filled out online from their homes at baseline and is a requirement to be able to participate in the study. At post intervention, and the three and six-month follow up participants will again receive an email asking them to fill out the questionnaires packet online using the link in the email. The data will be collected in a secure university approved system, RedCap. Follow-up emails, phone calls, and text message reminders will be sent out encouraging participants to fill out the surveys if they have not already done so.

Intervention:

CCT is an eight-week group based two-hour course and incorporates practices of compassion, mindfulness, and meditation, with scientific research on compassion and related topics in the fields of psychology and neurology along with contemplative thinking.

CCT is a psycho-educational course and each week participants engage with material on the cultivation of compassion and other related topics, class discussions, formal meditations, and dyadic exercises. Participants are asked to meditate daily at home for 20-25 minutes on guided compassion meditations accessed through the website www.centerforcompassion.dk and engage in informal compassion practices. The CCT course is curriculum-based and consists of 6 steps. Step 1 involves learning to focus and settle the mind. Step 2 involves cultivating the psychosomatic experiences of warmth and caring for a loved one. Step 3 involves training compassion and loving kindness for oneself. Step 4 involves cultivating compassion towards others through embracing our shared common humanity and appreciating the interconnectedness of self and others. Step 5 involves training compassion towards all beings, and step 6 involves an ''active compassion'' practice where participants imagine taking away others' pain and sorrow and offering them one's own joy and happiness (Jinpa, 2010).

Compliance and attrition Treatment compliance will be assessed by recording the number of completed CCT sessions, and by having participants fill out a daily practice log as research has shown that positive outcomes are dose dependent (Jazaieri et al., 2015). When applicable, participants will be asked for their reasons for poor compliance/drop-out and asked to continue participation in the assessments until six-months follow-up. Any adverse effects, reported by participants or observed by investigators, will be recorded and reported to the Research Ethics Committee (Duggan et al., 2014). An intention to treat (ITT) analysis will be used to circumvent noncompliance and missing outcomes, and to provide an unbiased estimate of treatment effects. When applicable, participants will be asked for their reasons for poor compliance/drop-out and asked to continue participation in the assessments until six-months follow-up.

Measures

Statistical Analysis:

We will compare the outcome variables (DASS, PSS, SCS-12, MCS, ERQ, BRS, FFMQ-15, and WHO-5) correcting for multiple comparisons where appropriate using the Student t or Wilcoxon tests. Analysis of covariance (ANCOVA) will be conducted to assess whether CCT is related to changes between baseline and after 8 weeks of intervention in relation to psychological distress.

The four measurement points allow to test whether changes in the proposed mediators are associated with changes in the proposed outcomes. This is a crucial condition in order to investigate mediators and possible mechanisms (Kazdin A.E., 2007). We will use structural equation modelling to examine the proposed mechanisms of CCT by testing the following action theories and conceptual theories simultaneously (Chen, H-T., 1994; Goldsmith et al., 2018).

The current project assumes two conceptual theories, which will be tested: 1) changes in compassion for self and others will affect psychological distress (DASS) and 2) changes in emotion regulation skills of reappraisal and suppression (ERQ) will affect psychological distress (DASS). The action theories, that CCT changes 1) compassion for self (SCS-12) and others (MCS) and 2) emotion regulation skills of reappraisal and suppression (ERQ), will be tested. The indirect, direct and total effects will be estimated with 95% CI inspired by a framework suggested by Goldsmith et al., (2018). The statistical package M-Plus will be applied.

We will also use a random-effects repeated measures analysis to examine the impact of the CCT intervention on psychological distress, adjusting for confounding variables (age, gender, ethnicity, socio-economic status, and years as informal caretaker). The repeated measure analysis approach accounts for the same individual's different outcome measures across different points in time without assuming either linear or curvilinear growth pattern. Cronbach alpha's will be computed to determine the internal consistency of our outcome measures.

Power:

The sample size was calculated using effect sizes from related publications (Jazaieri et al., 2013, 2014, 2015, Kuhlmann et al., 2015, Galante, et al., 2014, & Brito-Pons, 2014), respective η-square-values, and Cohen's d) with G*Power. The power analysis gave an approximate value of a minimum of 77 participants in both groups where we expect a medium effect size of .5 Cohen's d (alpha .05, power 80%). A minimum of 77 participants per group allows for an attrition rate of 20%, which will give us a minimum sample size of 64 participants per group. Four groups of approximately 20 participants per group will be given the CCT intervention.

Timeline 2018: Address the key points highlighted by the CCT participants who have taken the course (1-2 months). Ethics application has been approved (1 month). Recruitment of participants has begun (1 month -ongoing). A systematic review article: Mental health interventions for caregivers of people with mental illness: A systematic review and meta-analysis has been accepted by Prospero. (approved in July and will conclude in December 2018). Teach the first CCT course (20 participants) as part of the RCT in Southern Jutland (November -December 2018).

2019: Continue to deliver the main RCT (CCT versus wait list) intervention. Three CCT courses will be taught with approximately 20 participants in each class (January - April 2019). Begin collecting and interpreting data from participants (April - December 2019) and prepare second article: 'CCT for Caregivers: A randomized controlled trial' (November - December 2019).

2020: Collect and interpret final data from participants (January 2019), write dissertation and article on the main study. The article 'Compassion for Caregivers: Can compassion be utilized as an emotion regulation strategy in decreasing psychological distress?' (February - September 2020).

Research group:

Lone Fjorback (LF), Ph.D., MD is director of the Danish Mindfulness Centre, Institute of Clinical Medicine, Aarhus University with extensive expertise in clinical psychiatry and in constructing, advising and conducting high-quality research in the mindfulness field. Lone Fjorback is the main supervisor and principle investigator on this project.

Nanja Holland Hansen (NHH), cand.psych.aut and Ph.D.-student with Danish Center for Mindfulness, Institute of Clinical Medicine, Aarhus University, will carry out the intervention as she is a senior level CCT instructor. Nanja has extensive knowledge on compassion and compassion training. She was trained at Stanford University with some of the world's top experts in compassion and compassion training. She is also an experienced clinical psychologist and has worked nationally and internationally with a wide range of diverse populations and clinical issues.

Christine Parsons (CP), Ph.D. is an Associate Professor, with expertise in psychological science and neuroscience, from Interacting Minds Centre, Aarhus University and Oxford University. Christine has extensive knowledge regarding psychometric properties, statistical analysis and is a formidable researcher.

Lise Juul (LJ), Ph.D., is an Associate professor at Danish Center for Mindfulness, Institute of Clinical Medicine, Aarhus University. She has expertise in evaluating public health interventions and has conducted RCTs in real life settings and is highly competent within mediation analysis.

Karen-Johanne Pallesen (KJP) Ph.D., is an Associate Professor at the Danish Center for Mindfulness, Institute of Clinical Medicine, Aarhus University. Her expertise lies within the field of neuropsychology, cognitive science, and cognitive psychology.

On an advisory level, Leah Weiss (LW), PhD, a member of the founding faculty of the CCT program with the Compassion Institute, USA and Stanford University will collaborate on any CCT related issues, such as teaching concerns and CCT material.

Plan for dissemination Both positive and negative research results will be published in peer-reviewed journals, presented at international and national conferences and disseminated via media such as facebook, twitter, and the Danish Center for Mindfulness website. Knowledge about how to help informal caregivers and how to increase compassion will be shared with relevant organizations. The Danish Center for Mindfulness will continue to share the results that come out of the research. We already know, based on the pilot data, that the CCT course is feasible within a Danish context and for professional caregivers (i.e. doctors, psychologists, nurses etc.). These results have already been disseminated at two international conferences: The International Conference on Mindfulness, Amsterdam, Holland, Summer 2018, and Mind and Life Summer Research Institute, Germany, 2018.

Perspective The knowledge gained from this research will lead to a greater understanding of whether an 8-week compassion training course for informal caregivers is feasible but also the effect of the CCT course and possibility to ease the burden of being a caregiver. This is extremely important knowledge for implementation and improving current practice for informal caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. caregiver male and female (fx. parent /spouse/other family member) of a person with a mental illness,
2. 18 - 75 years of age
3. Danish speaking
4. not pregnant.

Exclusion Criteria:

1. having an untreated mental illness,
2. addictions, or substance abuse
3. meditation practice (studies have shown that people who are long-term meditation practitioners are more resilient and have greater psychological well-being (Lykins & Baer, 2009). Therefore, people with 1 year or more of prior formal meditation practice, will not be eligible for the study as we cannot rule out whether their scores are due to their long-term practice or to the CCT intervention),
4. or current psychotherapeutic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Change is being assessed: Depression Anxiety Stress Scales (DASS: Lovibond, S.H. & Lovibond, P.F., 1995) | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The DASS is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress.

SECONDARY OUTCOMES:
Change is being assessed: Perceived Stress Scale, (PSS: Cohen et al., 1983) | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The PSS assesses the perceived stress within the last month. It is a 14 item self-report questionnaire using a 5 point-likest scale.
Change is being assessed: The Emotion Regulation Questionnaire (ERQ: Gross & John, 2003). | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The ERQ is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: 1. Cognitive Reappraisal and 2. Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale.
Change is being assessed: Self-compassion Scale -12 (SCS-12: Raes et al., 2011). | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The SCS is a 12-item scale is designed to measure respondents level of self-compassion. Respondents answer on a 5-point Likert scale.
Change is being assessed: Multidimensional Compassion Scale (MCS: Jazaieri et al., 2018) | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The MCS scale is a general measure of compassion with four components: Cognitive, affective, intentional, and motivational. The scale is comprised of 16 questions and respondents answer on a 7-point Likert scale.
Change is being assessed: Five Facet Mindfulness Scale (FFMQ-15: Baer et al., 2006). | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The FFMQ is a 15-item scale measuring mindfulness. Respondents answer on a 5-point Likert Scale.
Change is being assessed: Brief Resilience Scale (BRS: Smith B. W. et al., 2008) | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The brief resilience scale (BRS) is a 6-item scale assessing the ability to bounce back or recover from stress.
Change is being assessed: Working Alliance Inventory Short Form Revised (WAI-SR: Horvath, A. O. et al (1989) & Tracey, T. J., & Kokotovic, A. M. (1989)). | week 2 and week 8 of the 8 week CCT program
  The WAI-SR is a 12-item scale measuring three domains of the therapeutic alliance: (a) agreement between patient and therapist on the goals of the treatment (Goal); (b) agreement between patient and therapist about the tasks to achieve these goals (Task); and (c) the quality of the bond between the patient and therapist (Bond). The WAI-SR is a patient-rated questionnaire. Patients rate items on a 5-point Likert scale
Change is being assessed: The World Health Organisation- Five Well-Being Index (WHO-5: Topp C.W. et al, 2015; Bech, P., 2012) | Baseline, 8 weeks, and 3-months and 6-months follow up.
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. The WHO-5 consists of five statements, which respondents rate according to the scale.

OTHER OUTCOMES:
Demographical questions | Baseline
  age, gender, income, educational status, years of informal caregiving

CONTACTS AND LOCATIONS:
Overall Officials: Lone Fjorback, MD, Study Director — Aarhus University, Danish Center for mindfulness
Locations (2):
- Denmark (2):
  - Aarhus Universitet, Copenhagen
  - Aarhus University, Kolding

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jinpa, T. (2010). Compassion cultivation training program (CCT program): An eight-week course on cultivation a compassionate heart and mindset. Instructor's Manual. The Center for Compassion and Altruism Research and Education (CCARE). Stanford Institute for Neuro-Innovation and Translational Neuroscience, Stanford University (Unpublished).
- [Background] Jazaieri, H., Lee, I.A., McGonigal, K., Jinpa, T., Doty, J.R., Gross, J.J., & Goldin, P.R.,(2015). A wandering mind is a less caring mind: Daily experience sampling during compassion meditation training. The Journal of Positive Psychology, Routledge
- [Background] Duggan C, Parry G, McMurran M, Davidson K, Dennis J. The recording of adverse events from psychological treatments in clinical trials: evidence from a review of NIHR-funded trials. Trials. 2014 Aug 27;15:335. doi: 10.1186/1745-6215-15-335. PMID 25158932
- [Background] Kazdin AE. Mediators and mechanisms of change in psychotherapy research. Annu Rev Clin Psychol. 2007;3:1-27. doi: 10.1146/annurev.clinpsy.3.022806.091432. PMID 17716046
- [Background] Chen, H-T., (1994). Theory-driven evaluations: Need, difficulties, and option. American Journal of Evaluations, 15, pp. 79-82.
- [Background] Goldsmith KA, MacKinnon DP, Chalder T, White PD, Sharpe M, Pickles A. Tutorial: The practical application of longitudinal structural equation mediation models in clinical trials. Psychol Methods. 2018 Jun;23(2):191-207. doi: 10.1037/met0000154. Epub 2017 Dec 28. PMID 29283590
- [Background] Jazaieri, H., Jinpa, T., McGonigal, K., Rosenberg, E., Finkelstein, J., Simon-Thomas, E., & Goldin, P.R. (2013). Enhancing compassion: randomized controlled trial of a compassion cultivation training program. Journal of Happiness Studies, 14, pp. 1113-1126.
- [Background] Kuhlmann SM, Burger A, Esser G, Hammerle F. A mindfulness-based stress prevention training for medical students (MediMind): study protocol for a randomized controlled trial. Trials. 2015 Feb 8;16:40. doi: 10.1186/s13063-014-0533-9. PMID 25887430
- [Background] Galante J, Galante I, Bekkers MJ, Gallacher J. Effect of kindness-based meditation on health and well-being: a systematic review and meta-analysis. J Consult Clin Psychol. 2014 Dec;82(6):1101-14. doi: 10.1037/a0037249. Epub 2014 Jun 30. PMID 24979314
- [Background] Brito, G.P. (2014). Cultivating healthy minds and open hearts. A mixed method controlled study on the psychological effects of compassion cultivation training in Chile. A dissertation submitted in partial fulfillment of the requirements for the degree of Doctor of Philosophy in transpersonal psychology, Sofia University, Palo Alto, California, USA.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Jazaieri, H., McGonigal, K., Jinpa, T., Doty, J.R., Gross, J.J., & Goldin, P.R. (2014). A randomized controlled trial of compassion cultivation training: Effects on mindfulness, affect, and emotion regulation. Motivation and Emotion, 38, pp. 23-35
- [Background] Jazaieri, H., Lee, I.A., McGonigal, K., Jinpa, T., Doty, J.R., Gross, J.J., & Goldin, P.R.,(2015). A wandering mind is a less caring mind: Daily experience sampling during compassion meditation training. The Journal of Positive Psychology, Routledge.
- [Background] Jazaieri, H., Goldin, P. R., Simon-Thomas, E., Keltner, D., & Mendoza-Denton, R. (in prep). Predicting Compassionate Behavior: Application, development, and psychometric properties of the Multidimensional Compassion Scale.
- [Background] Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety Stress Scales. (2nd. Ed.) Sydney: Psychology Foundation. ISBN 7334-1423-0.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Horvath, Adam O.,Greenberg, Leslie S. (1989). Development and validation of the Working Alliance Inventory.Journal of Counseling Psychology, Vol 36(2), Apr 1989, 223-233
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Lykins, E.R.B., & Baer, R.A. (2009). Psychological functioning in a sample of longtern practioners of mindfulness meditation. Journal of Cognitive Psychotherapy, 23, (3), pp. 226-241.
- [Background] Bech P. (2012). Clinical Psychometrics , Wiley-Blackwell, Oxford.
- [Background] Tracey, T. J., & Kokotovic, A. M. (1989). Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology, 1(3), 207-210.
- [Derived] Hansen NH, Juul L, Pallesen KJ, Fjorback LO. Effect of a Compassion Cultivation Training Program for Caregivers of People With Mental Illness in Denmark: A Randomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e211020. doi: 10.1001/jamanetworkopen.2021.1020. PMID 33683334